CLINICAL TRIAL: NCT01802905
Title: Utilization of Genomic Information to Augment Chemotherapy Decision-making for People With Incurable Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: BC Cancer Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: BCCA POG 01
Record Dates: First submitted 2013-02-27; First posted 2013-03-04 (Estimated); Last update posted 2015-02-05 (Estimated); Status verified 2013-02

CONDITIONS: Advanced Incurable Cancers
Keywords: neoplasm; metastatic cancer; cancer genome; genomic analysis; adults
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sequenced patients (Experimental): Patients enrolled on the study who have successful sequencing of their cancers will be closely monitored for: what chemotherapy agents are next used, what response and toxicity do they have, is there any early sign of response detected on PET-CT, overall did the genomic information change treatment decision-making.
  Interventions: Genetic: in depth genomic sequencing

INTERVENTIONS:
Genetic: in depth genomic sequencing — Fresh tumour biopsies and matched normal specimens (blood and surrounding tissue) and when possible archival pretreatment specimens, will undergo in depth DNA and RNA sequencing and analysis on an oncogene panel.

SUMMARY:
Most systemic therapies are chosen on the basis of large randomized clinical trials; however, tumour heterogeneity means that cancers with similar histological features may have substantially different underlying biological drivers. The investigators propose that applying personal genomic information prospectively obtained in a clinically realistic timeframe to assist in chemotherapy decision-making could result in more effective and efficient cancer treatment. This study will investigate this approach in a cross section of advanced cancers to examine timeliness, deliverability, rate of actionable targets identified, and our ability to expand this approach into a larger clinical trial setting.

DETAILED DESCRIPTION:
It is clear that carcinogenesis is an immensely complex process and that even within a histologic cancer subtype - such as adenocarcinoma of the lung or breast - there is significant heterogeneity in cancer behaviour and response to therapy. Recognizing genetic mutations that promote disease facilitates targeted treatment; this has been demonstrated in several small subgroups of cancers in which specific genetic mutations or translocations have been successfully treated with targeted chemotherapy agents.

Analyses of individual patients demonstrate unique molecular signatures for every cancer examined. Frequently, multiple different pathways are involved in disease growth and progression and the dominant process varies from person to person and perhaps even within different sites of disease within one person. As well these variations evolve in response to treatment. With many recognized mutations personalized evaluation of the genetic signature encoded in DNA and RNA may enable directed therapy to the appropriate oncologic pathway thereby providing information to help guide chemotherapy choices.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must have histologically or cytologically confirmed diagnosis of cancer
2. This cancer must be incurable, as defined by their treating oncologist (generally because of advanced stage).
3. Subjects must agree to provide archival tissue and agree to undergo a study specific biopsy and blood test for genetic analysis. All subjects would have a biopsy and blood samples at progression if it could be done safely.
4. ECOG PS 0 or 1.
5. Age > 18 years of age.
6. Subject consent must be obtained according to the BCCA requirements.
7. Subject must be accessible for treatment and follow-up. Subjects must be registered at the BCCA Vancouver site.

Exclusion Criteria:

1. Unable or unwilling to undergo tumour biopsy(s) and/or blood/skin samples for normal DNA.
2. Significant medical condition that in the opinion of the treating oncologist renders the subject not suitable for participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Frequency of actioanble genomic abnormalites detected that modify treatment | up to 24 months
  What is the frequency of "actionable" results in this varied tumour population ?

SECONDARY OUTCOMES:
What is the frequency with which these actionable results actually result in a subject receiving a drug(s) related to this test | up to 24 months
  What is the frequency with which these actionable results actually result in a subject receiving a drug(s) related to this test.

CONTACTS AND LOCATIONS:
Overall Officials: Janessa J. Laskin, MD FRCPC, Principal Investigator — British Columbia Cancer Agency; Marco Marra, PhD FRSC, Principal Investigator — Genome Sciences Centre, BC Cancer Agency
Locations (1):
- BC Cancer Agency, Vancouver, British Columbia, Canada

REFERENCES:
- [Background] Peixoto RD; Li Y; Pleasance E; Yip S; et al. A case of the utilization of genomic information in the management of metastatic colorectal cancer. J Clin Oncol 30: 2012 (suppl 34; abstr 444)